CLINICAL TRIAL: NCT04195672
Title: Official Title Evaluation of the Value of Newborn Infant Parasympathetic Evaluation (NIPE) in Sedated/Ventilated Patients in Pediatric Intensive Care Unit
Brief Title: NIPE as an Indicator of Pain in Sedated/Ventilated Patient Under 3 Years-old Hospitalized in Intensive Care Unit
Acronym: NIPE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: NI2019_
Record Dates: First submitted 2019-12-02; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Ventilator Lung; Newborn
Keywords: Pediatric; Pain; Heart rate variability; Intensive care unit; Analgesia
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children under 3 years-old intubated/sedated in intensive care: NIPE and CBS ware measured for each included patient
  Interventions: Device: NIPE (MDoloris®) and CBS values

INTERVENTIONS:
Device: NIPE (MDoloris®) and CBS values — During different procedures of care with the bed-side nurse, NIPE ware recorded. Monitoring started 15 minutes before care and continuously recorded until 10 minutes after the procedure. Pain assessment was evaluated by the CBS under 3 periods for each patient: 1- before any procedure (T1) representing the baseline, 2- during the procedure of care (T2), and 3- after the procedure (T3). Investigator who performed the CBS was blind to NIPE during the procedure recording.
  This study did not change the procedure of care before or after and had no impact on care

SUMMARY:
The main objective is to assess correlation between Newborn Infant Parasympathetic Index values and external evaluation by Comfort Behaviour Scale during painful medical cares in sedated intubated children admitted in pediatric intensive care unit.

DETAILED DESCRIPTION:
The assessment of pain in patient hospitalized in intensive care remains a challenge, especially for patients which are unable to communicate their pain intensity. Self-reported scales are widely used for children's pain assessment but cannot be used in sedated or non-communicable patients. The gold standard for pain evaluation in sedated-ventilated patient in pediatric intensive care unit is the Comfort Behaviour Scale (CBS). However, this method remains subjective, depending on training and ability to use this clinical tool by the examiner. The Newborn Infant Parasympathetic Evaluation (NIPE) is a non-invasive system based on the analysis variability in high frequency (> 0.15 Hz) which reflects the parasympathetic activity related to respiratory fluctuations of heart rate. With a numerical index ranging from 0 to 100, NIPE values, measured continuously, has been developed to evaluate the degree of pain intensity. In this study, the hypothese is the NIPE could be used as an indicator of pain in sedated/intubated children under 3 years-old hospitalized in Pediatric intensive care unit.

This study did not change the procedure of care before or after and had no impact on care.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patient ≤ 3 year-old, mechanically ventilated

Exclusion Criteria:

* Withdraw life-support,
* unstable condition preventing planned routine procedures of care,
* conditions precluding the use of NIPE (cardiac transplant, absence of sinus cardiac rhythm, apnea or respiratory rate ≤ 25 /min, pacemaker and use of atropine and/or isoprenaline and conditions of days of availability for NIPE)

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All consecutive patient ≤ 3 year-old, mechanically ventilated
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Newborn Infant Parasympathetic Evaluation | Through the study completion (18 months)
  Comparison between Newborn Infant Parasympathetic Evaluation values (0 to 100) and Comfort Behaviour Scale values (8 to 40) assessed by coefficient of correlation in patients upper than three years old
Comfort Behaviour Scale | Through the study completion (18 months)
  Comparison between Newborn Infant Parasympathetic Evaluation values (0 to 100) and Comfort Behaviour Scale values (8 to 40) assessed by coefficient of correlation in patients upper than three years old

SECONDARY OUTCOMES:
Newborn Infant Parasympathetic Evaluation | Through the study completion (18 months)
  Determination of pain detection threshold with Newborn Infant Parasympathetic Evaluation scale (0 to 100) using receiving operator characteristics (ROC) curve

CONTACTS AND LOCATIONS:
Overall Officials: morgan Recher, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHU, Lille, France

REFERENCES:
- [Derived] Recher M, Rousseaux J, Flocteil M, Jouancastay M, Potisek A, Lampin ME, Leteurtre S, De Jonckheere J. Assessment of Procedural Distress in Sedated/Intubated Children Under 3 Years Old Using the Newborn Infant Parasympathetic Evaluation: A Diagnostic Accuracy Pilot Study. Pediatr Crit Care Med. 2020 Dec;21(12):e1052-e1060. doi: 10.1097/PCC.0000000000002454. PMID 32740184